CLINICAL TRIAL: NCT06132087
Title: PROACTIVE Pilot Study: Pancreatic Resection Outcomes in Locally Advanced Pancreatic Cancer Involving Visceral Arteries Treated With Neoadjuvant Chemotherapy
Brief Title: PROACTIVE: Surgical Resection Outcomes in Locally Advanced and Unresectable Pancreatic Cancer After Neoadjuvant Chemotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3P-23-5; NCI-2023-09210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3P-23-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer American Joint Committee on Cancer v8; Unresectable Pancreatic Adenocarcinoma
MeSH Terms: interventions — Specimen Handling; Laparoscopy; Magnetic Resonance Spectroscopy; Pancreaticoduodenectomy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (surgical resection) (Experimental): Patients undergo laparoscopy followed by surgical resection with pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy at the discretion of the surgeon within 2-8 weeks following completion of standard of care neoadjuvant chemotherapy regimen. Patients undergo CT and blood sample collection throughout the study and/or MRI during screening. Patients also undergo tissue collection at time of surgical resection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Distal Pancreatectomy; Procedure: Laparoscopy; Procedure: Magnetic Resonance Imaging; Procedure: Pancreaticoduodenectomy; Other: Questionnaire Administration; Procedure: Surgical Procedure; Procedure: Total Pancreatectomy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; Computed Axial Tomography (CAT); Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Distal Pancreatectomy — Undergo distal pancreatectomy
Procedure: Laparoscopy — Undergo laparoscopy
  Other Names: Peritoneoscopy; Keyhole surgery
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; Nuclear Magnetic Resonance Imaging (NMRI); Nuclear Magnetic Resonance
Procedure: Pancreaticoduodenectomy — Undergo pancreaticoduodenectomy
  Other Names: Pancreatoduodenectomy
Other: Questionnaire Administration — Ancillary studies
Procedure: Surgical Procedure — Undergo surgical resection
  Other Names: Operation; Surgery; Surgery Type; Surgery, Not Otherwise Specified; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
Procedure: Total Pancreatectomy — Undergo total pancreatectomy
  Other Names: Total Excision of the Pancreas

SUMMARY:
This clinical trial tests how well surgical resection after chemotherapy given before surgery to make the tumor smaller (neoadjuvant) works to treat pancreatic cancer that has spread to nearby tissue or lymph nodes (locally advanced) and that cannot be removed by surgery (unresectable). In general, surgery is considered the most effective treatment for pancreatic cancer, especially when the cancer is localized and has not spread to other organs. However, most patients with pancreatic cancer are not candidates for surgical removal because the cancer has grown into or close to nearby arteries, veins, or organs and there is a concern of damaging these nearby structures. Researchers want to find out if surgery after neoadjuvant chemotherapy can be done safely to completely remove the tumor in patients with locally advanced and unresectable pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the R0 resection in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

SECONDARY OBJECTIVES:

I. To evaluate overall survival (OS) in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

II. To measure disease free survival (DFS) in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

III. To evaluate the correlation between post-neoadjuvant/preoperative radiological staging and pathologic staging.

IV. To estimate time to distant metastases (TDM) in patients in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation between post-neoadjuvant/preoperative radiological staging and pathologic staging.

II. To evaluate objective response rate (ORR) in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy.

III. To assess if mutations on next-generation sequencing (NGS) testing and the change in circulating tumor deoxyribonucleic acid (ctDNA) pre- and post-operative is predictive of DFS or OS in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

IV. To evaluate the rate of unresectability in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy.

V. To evaluate pathologic tumor response and rate of pathologic complete response (pCR) in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

VI. To evaluate correlation between R0 resection rate and pathologic treatment response and survival outcomes.

VII. To evaluate number of cycles of perioperative chemotherapy received in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

VIII. To evaluate the adverse event profile in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

IX. To evaluate the physical functioning, nausea/vomiting, and diarrhea, as measured with the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire 30 (EORTC QLQ-C30) in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

X. To evaluate the average operative time in minutes in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

XI. To evaluate the estimated blood loss (mL) in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

XII. To assess the length of hospital, stay in for patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

XIII. To evaluate the incidence of thrombosis in patients with locally advanced pancreatic adenocarcinoma treated with perioperative chemotherapy and surgery.

OUTLINE:

Patients undergo laparoscopy followed by surgical resection with pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy at the discretion of the surgeon within 2-8 weeks following completion of standard of care neoadjuvant chemotherapy regimen. Patients undergo computed tomography (CT) and blood sample collection throughout the study and/or magnetic resonance imaging (MRI) during screening. Patients also undergo tissue collection at time of surgical resection on study.

After completion of study intervention, patients are followed up at 30 days, every 3 months for the first year, then every 6 months until 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic proof of pancreatic adenocarcinoma
* Locally advanced, stage III (T4NxM0) and unresectable by National Comprehensive Cancer Network (NCCN) Guidelines prior to perioperative chemotherapy
* Patients must have measurable disease at diagnosis per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* At least 4 cycles of perioperative chemotherapy (gemcitabine [Gem]/nab-paclitaxel or fluorouracil, irinotecan, leucovorin and oxaliplatin [FOLFIRINOX]) received with no evidence of progression on restaging scans per RECIST 1.1
* Age ≥ 18 years
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-1
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcl
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) if no biliary stenting has been done or 2.0 x ULN if patient is status post (s/p) biliary stenting or two down trending values
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase [SPGT]) ≤ 2.5 X ULN
* Creatinine (Cr) ≤ 1.5 mg/dL or Cr clearance ≥ 30 mL/min (as estimated by Cockcroft Gault)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patient with known distant metastases
* Patients who have not recovered from adverse events of chemotherapy due to agents administered more than 4 weeks earlier
* Patients who have progressed on 2 prior systemic chemotherapy lines or received prior radiotherapy for pancreatic cancer
* Patients may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | At time of surgery
  Will be defined as the proportion of patients with negative resection margins after undergoing surgery.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Determined from the date of registration to the date of death due to any cause.
Disease-free survival | Up to 2 years
  Determined from the date of registration to the date of progression prior to surgery, metastases detected during surgery, recurrence (locoregional and/or distant) after resection, and death due to any cause, whichever occurs first.
Time to locoregional recurrence | Up to 2 years
  Determined from the date of registration to the date of locoregional recurrence after resection.
Time to distant metastases | Up to 2 years
  Determined from the date of registration to the date of metastases prior to surgery, metastases detected during surgery, or distant recurrence after resection.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Grossman, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States